CLINICAL TRIAL: NCT02509767
Title: Depo Provera Self-Administration Study: Putting a Patient-Centered Practice to the Test at Planned Parenthood
Acronym: DSAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Planned Parenthood Federation of America (Other)
Collaborators: Pfizer (Industry); Tara Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00012433; DSAS-2015 (Other: Planned Parenthood Federation of America)
Record Dates: First submitted 2015-07-25; First posted 2015-07-28 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Contraception
Keywords: Contraceptive Methods; Female Contraception; Contraceptive satisfaction; Injectable contraception; Birth control
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Administration (Experimental): Subjects who are randomized to self-administration will be taught self-administration of subcutaneous depot medroxyprogesterone acetate (DMPA sc) by a clinic nurse or other qualified personnel using instructions based on the packaging insert. If willing, subjects will then self-administer DMPA sc under supervision. Subjects who are able to correctly self-administer DMPA sc as assessed by the supervising nurse and who are interested in continued home self-administration will then be provided medication (3 doses of DMPA sc), a self-administration kit (includes alcohol swabs, cotton pads, bandages, mini sharps disposal container), and instructions to do so for the subsequent 3 injections indicating the appropriate dates for injection. All subjects will receive reminders when their next injection is due.
  Interventions: Drug: Subcutaneous depot medroxyprogesterone acetate
- Clinic Administration (Standard Care) (Other): Subjects who are randomized to clinic administration will receive subcutaneous depot medroxyprogesterone acetate (DMPA sc) injection administered by a clinic nurse or other qualified personnel and receive standard care. They will be instructed to make an appointment to return to the clinic as usual to receive subsequent injections every 12-14 weeks. All subjects will receive reminders when their next injection is due.
  Interventions: Drug: Subcutaneous depot medroxyprogesterone acetate

INTERVENTIONS:
Drug: Subcutaneous depot medroxyprogesterone acetate — Based on study arm, subjects will either be taught to self-inject or will be administered DMPA sc by qualified clinic personnel.
  Other Names: depo-subQ provera 104™

SUMMARY:
This randomized clinical trial will study subcutaneous depot medroxyprogesterone acetate (DMPA sc) self-administration at two Planned Parenthood affiliates serving diverse patient populations. Prior studies demonstrate that DMPA self-injection is safe, effective, feasible, and acceptable for women and adolescents. A total of 400 female patients (ages 15-44) requesting DMPA will be randomized to self-administration of DMPA sc or clinic administration (usual care). Subjects will be followed for one year. The primary study outcome is DMPA continuation at one year by self-report in both study arms. Secondary outcomes include patient-reported satisfaction with treatment; satisfaction with home use; and costs associated with contraceptive care. The investigators hypothesize higher continuation rates among self-injection users compared to patients who receive standard care. Secondary exploratory hypotheses include higher patient satisfaction and lower costs associated with contraceptive care among self-injection users.

DETAILED DESCRIPTION:
This open-label, randomized parallel group clinical trial will study subcutaneous depot medroxyprogesterone acetate (DMPA sc) self-administration at two Planned Parenthood affiliates serving diverse patient populations. Prior studies demonstrate that DMPA self-injection is safe, effective, feasible, and acceptable for women and adolescents. A total of 400 female patients (ages 15-44) requesting DMPA will be randomized to self-administration of DMPA sc or clinic administration (usual care) in a 1:1 allocation. Subjects will be followed for one year. All subjects will receive reminders when their next injection is due. Follow-up surveys will be conducted at 6 and 12 months. Adherence will be monitored by subject self-report and study outcomes will be ascertained by self-report and medical record review.

The primary study outcome is DMPA continuation at one year by self-report in both study arms. Secondary outcomes include patient-reported satisfaction with treatment; satisfaction with home use; and costs associated with contraceptive care.

The investigators hypothesize higher continuation rates among self-injection users compared to patients who receive standard care (delta = .13; 80% power; one-sided α=0.05; allowing for 15% loss-to-follow-up). Secondary exploratory hypotheses include higher patient satisfaction and lower costs associated with contraceptive care among self-injection users.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 15-44
* Current or past users of DMPA or desires initiation of DMPA for contraception
* Can understand spoken and written English or Spanish
* Willing to consider/attempt DMPA self-injection
* Willing to be randomized to either self- or clinic administration of DMPA
* Do not want to become pregnant in the next 12 months
* Willing to provide contact information and to complete three surveys at baseline, 6 months, and 12 months
* Have consistent access to a working telephone, email, and Internet
* No contraindications to DMPA use

Exclusion Criteria:

* Suspected or confirmed pregnancy
* Vaginal bleeding of unknown etiology
* Known or suspected breast cancer
* Acute liver disease
* High blood pressure (Systolic ≥ 160 mm Hg or diastolic ≥ 100 mm Hg)
* Known hypersensitivity to medroxyprogesterone acetate or any other components of DMPA
* Desire for pregnancy within one year

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 401 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia E Kohn, PhD, MPA, Principal Investigator — Planned Parenthood Federation of America
Locations (2):
- United States (2):
  - Planned Parenthood of Central and Greater Northern New Jersey, Morristown, New Jersey
  - Planned Parenthood Gulf Coast, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-Administration | Clinic Administration (Standard Care)
Started | 201 | 200
Completed | 157 | 159
Not Completed | 44 | 41

BASELINE CHARACTERISTICS:
Population: One subject who was randomized to the self-administration arm enrolled and immediately withdrew from the study. Therefore the total number enrolled was 401, but the total number analyzed was 400.
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Administration | Clinic Administration (Standard Care) | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (6.5) | 26.0 (6.2) | 26.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject randomized to the self-administration group enrolled and then immediately withdrew from the study. Therefore a total of 401 subjects were enrolled (201 in the self-administration arm and 200 in the clinic administration arm), but only 400 were included in the analysis population (200 in each study arm).
  Participants
    Female | 200 | 200 | 400
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Hispanic | 98 | 106 | 204
  Race/ethnicity: Non-Hispanic White | 40 | 31 | 71
  Race/ethnicity: Non-Hispanic Black | 56 | 51 | 107
  Race/ethnicity: Asian / Pacific Islander | 2 | 6 | 8
  Race/ethnicity: Other | 1 | 6 | 7
  Race/ethnicity: Unknown | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Northeast | 100 | 100 | 200
  United States: South | 100 | 100 | 200
DMPA user status at enrollment [Count of Participants; unit: Participants]
  Current DMPA user | 83 | 88 | 171
  Past DMPA user | 27 | 26 | 53
  New DMPA user | 89 | 85 | 174
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Depot Medroxyprogesterone Acetate (DMPA sc) Continuation at One Year by Self-report in Both the Self- and Clinic Administration Arms
Description: Number of participants with Depot Medroxyprogesterone Acetate (DMPA sc) continuation at one year by self-report in both the self- and clinic administration arms measured by self-administered questionnaire.
Time Frame: 12 months from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Administration | Clinic Administration (Standard Care)
Number analyzed (Participants) | 157 | 159
Participants | 108 | 85

2. Secondary Outcome: Number of Participants Who Were Satisfied With Depot Medroxyprogesterone Acetate (DMPA sc) at One Year by Self-Report in Both the Self- and Clinic Administration Arms
Description: Number of participants who reported being very or somewhat satisfied with Depot Medroxyprogesterone Acetate (DMPA sc) at one year in both the self- and clinic administration arms measured by self-administered questionnaire.
Time Frame: 12 months from enrollment
Population: Analysis population only includes participants who had complete outcome data for both the 6- and 12-month surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinic Administration (Standard Care) | Self-Administration
Number analyzed (Participants) | 159 | 157
Participants | 147 | 137

3. Secondary Outcome: Number of Participants Who Were Satisfied With Home Use of Depot Medroxyprogesterone Acetate (DMPA sc) at One Year by Self-Report in the Self-Administration Arm
Description: Number of participants who were satisfied with home use of Depot Medroxyprogesterone Acetate (DMPA sc) at one year by self-report in the self-administration arm only as measured by self-administered questionnaire.
Time Frame: 12 months from enrollment
Population: Analysis population only includes participants who had complete outcome data for both the 6- and 12-month surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Administration
Number analyzed (Participants) | 157
Participants | 137

4. Secondary Outcome: Costs Associated With Contraceptive Care
Description: Costs associated with contraceptive care measured by self-administered questionnaire.
Time Frame: 6 and 12 months from enrollment
Population: We did not collect the data necessary to ascertain results for this outcome. While this was originally planned as a secondary study outcome, we utlimately determined that it was not feasible. Therefore we have reported "0" for this outcome and are unable to report results.
Arm/Group | Self-Administration | Clinic Administration (Standard Care)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected for subjects for a period of 1 year following study enrollment (i.e. baseline).
Arm/Group | Self-Administration | Clinic Administration (Standard Care)
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/201 | 0/200
Other Adverse Events (participants affected / at risk) | 0/201 | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT02509767/Prot_SAP_000.pdf